CLINICAL TRIAL: NCT02448368
Title: A Phase 1, Randomized, Open-Label, Study in Healthy Adult Male Subjects to Assess the Relative Bioavailability and Food Effect of Various Formulations of RDEA3170
Brief Title: RDEA3170 Tablet and Capsule Bioavailability Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RDEA3170-111
Record Dates: First submitted 2015-04-30; First posted 2015-05-19 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2017-11

CONDITIONS: Healthy
MeSH Terms: interventions — verinurad

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Treatment A (Experimental): RDEA3170, 5 mg (FN24), administered in the fasted state.
  Interventions: Drug: RDEA3170, 5 mg
- Treatment B (Experimental): RDEA3170, 5 mg (FN24), administered in the fed state (high-fat, high-calorie meal).
  Interventions: Drug: RDEA3170, 5 mg
- Treatment C (Experimental): RDEA3170, 10 mg (FN25), administered in the fasted state.
  Interventions: Drug: RDEA3170,10 mg
- Treatment D (Experimental): RDEA3170, 10 mg (FN25), administered in the fed state (high-fat, high-calorie meal).
  Interventions: Drug: RDEA3170,10 mg
- Treatment E (Experimental): RDEA3170, 2.5 mg (FN17), administered as 10 mg (4 × 2.5 mg), in the fasted state.
  Interventions: Drug: RDEA3170, 2.5 mg
- Treatment I (Experimental): RDEA3170, 10 mg (FN26), administered in the fasted state.
  Interventions: Drug: RDEA3170, 10 mg
- Treatment J (Experimental): RDEA3170, 10 mg (FN26), administered in the fed state (high-fat, high-calorie meal).
  Interventions: Drug: RDEA3170, 10 mg
- Treatment K (Experimental): RDEA3170, 2.5 mg (FN17), administered as 10 mg (4 × 2.5 mg), in the fasted state.
  Interventions: Drug: RDEA3170, 2.5 mg

INTERVENTIONS:
Drug: RDEA3170,10 mg — Approximately 20 subjects will be randomized to 1 of 10 treatment sequences with single doses occurring on Days 1, 5, 9, 13, and 17.
  Other Names: Cohort 1
  Arms: Treatment C; Treatment D
Drug: RDEA3170, 2.5 mg — Approximately 20 subjects will be randomized to 1 of 10 treatment sequences with single doses occurring on Days 1, 5, 9, 13, and 17.
  Other Names: Cohort 1
  Arms: Treatment E
Drug: RDEA3170, 5 mg — Approximately 20 subjects will be randomized to 1 of 10 treatment sequences with single doses occurring on Days 1, 5, 9, 13, and 17.
  Other Names: Cohort 1
  Arms: Treatment A; Treatment B
Drug: RDEA3170, 10 mg — Fifteen subjects were randomized to 1 of 3 treatment sequences with single doses occurring on Days 1, 5, and 9.
  Other Names: Cohort 3
  Arms: Treatment I; Treatment J
Drug: RDEA3170, 2.5 mg — Fifteen subjects were randomized to 1 of 3 treatment sequences with single doses occurring on Days 1, 5, and 9.
  Other Names: Cohort 3
  Arms: Treatment K

SUMMARY:
The purpose of this study is to determine the relative bioavailability of RDEA3170 capsules compared with RDEA3170 tablets.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the study procedures and the risks involved, and is willing to provide written informed consent before the first study-related activity.
* Subject has a body weight ≥ 50 kg (110 lbs.) and a body mass index ≥ 18 and ≤ 40 kg/m2.
* Subject has a Screening serum urate level of 4 to 7 mg/dL.
* Subject is free of any clinically significant disease or medical condition, per the Investigator's judgment.

Exclusion Criteria:

* Subject has a history or suspicion of kidney stones.
* Subject has undergone major surgery within 3 months prior to Screening.
* Subject donated blood or experienced significant blood loss within 12 weeks prior to Day 1 or gave a plasma donation within 4 weeks prior to Day 1.
* Subject has clinically unacceptable physical examination, per the Investigator's judgment.
* Subject has clinically relevant abnormalities in blood pressure, heart rate, or body temperature, per the Investigator's judgment.
* Subject has Screening clinical safety laboratory parameters (serum chemistry [other than serum creatinine and serum urate], hematology, coagulation or urinalysis) that are outside the normal limits and are considered clinically significant by the Investigator.
* Subject has a serum creatinine value above the upper limit of normal at the Screening visit.
* Subject has clinically relevant abnormalities in 12-lead electrocardiogram, per the Investigator's judgment.
* Subject has a history of cardiac abnormalities
* Subject cannot swallow multiple tablets or capsules.
* Subject has received any strong or moderate enzyme-inducing drug or product within 2 months prior to Day 1.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2015-06-26 (Actual); Study Completion 2016-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Hall, MD, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 35 participants were randomized
Pre-assignment Details: Twenty subjects were randomized to 1 of 10 treatment sequences in Cohort 1 with single doses. Fifteen subjects were randomized to 1 of 3 treatment sequences (IJK, JKI, and KIJ) in optional Cohort 3, with single doses occurring on Days 1, 5, and 9. The optional Cohort 2 to evaluate RDEA3170 capsules, 5 mg FN23 was not conducted per Sponsor decision.
Groups:
- Cohort 1: Sequence ABECD (Days 1, 5, 9, 13, and 17): 5 mg FN24 capsules, fasted; 5 mg FN24 capsules, fed; 10 mg FN17 tablets, fasted; 10 mg FN25 capsules, fasted; 10 mg FN25 capsules, fed
- Cohort 1: Sequence AEBDC (Days 1, 5, 9, 13, and 17): 5 mg FN24 capsules, fasted; 10 mg FN17 tablets, fasted; 5 mg FN24 capsules, fed; 10 mg FN25 capsules, fed; 10 mg FN25 capsules, fasted
- Cohort 1: Sequence EADBC (Days 1, 5, 9, 13, and 17): 10 mg FN17 tablets, fasted; 5 mg FN24 capsules, fasted; 10 mg FN25 capsules, fed; 5 mg FN24 capsules, fed; 10 mg FN25 capsules, fasted
- Cohort 1: Sequence EDACB (Days 1, 5, 9, 13, and 17): 10 mg FN17 tablets, fasted; 10 mg FN25 capsules, fed; 5 mg FN24 capsules, fasted; 10 mg FN25 capsules, fasted; 5 mg FN24 capsules, fed
- Cohort 1: Sequence DECAB (Days 1, 5, 9, 13, and 17): 10 mg FN25 capsules, fed; 10 mg FN17 tablets, fasted; 10 mg FN25 capsules, fasted; 5 mg FN24 capsules, fasted; 5 mg FN24 capsules, fed
- Cohort 1: Sequence BACED (Days 1, 5, 9, 13, and 17): 5 mg FN24 capsules, fed; 5 mg FN24 capsules, fasted; 10 mg FN25 capsules, fasted; 10 mg FN17 tablets, fasted; 10 mg FN25 capsules, fed
- Cohort 1: Sequence BCADE (Days 1, 5, 9, 13, and 17): 5 mg FN24 capsules, fed; 10 mg FN25 capsules, fasted; 5 mg FN24 capsules, fasted; 10 mg FN25 capsules, fed; 10 mg FN17 tablets, fasted
- Cohort 1: Sequence CBDAE (Days 1, 5, 9, 13, and 17): 10 mg FN25 capsules, fasted; 5 mg FN24 capsules, fed; 10 mg FN25 capsules, fed; 5 mg FN24 capsules, fasted; 10 mg FN17 tablets, fasted
- Cohort 1: Sequence CDBEA (Days 1, 5, 9, 13, and 17): 10 mg FN25 capsules, fasted; 10 mg FN25 capsules, fed; 5 mg FN24 capsules, fed; 10 mg FN17 tablets, fasted; 5 mg FN24 capsules, fasted
- Cohort 1: Sequence DCEBA (Days 1, 5, 9, 13, and 17): 10 mg FN25 capsules, fed; 10 mg FN25 capsules, fasted; 10 mg FN17 tablets, fasted; 5 mg FN24 capsules, fed; 5 mg FN24 capsules, fasted
- Cohort 3: Sequence IJK (Days 1, 5, and 9): 10 mg FN26 capsules, fasted; 10 mg FN26 capsules, fed; 10 mg FN17 tablets, fasted
- Cohort 3: Sequence JKI (Days 1, 5, and 9): 10 mg FN26 capsules, fed; 10 mg FN17 tablets, fasted; 10 mg FN26 capsules, fasted
- Cohort 3: Sequence KIJ (Days 1, 5, and 9): 10 mg FN17 tablets, fasted; 10 mg FN26 capsules, fasted; 10 mg FN26 capsules, fed
Period: Overall Study
Arm/Group | Cohort 1: Sequence ABECD (Days 1, 5, 9, 13, and 17) | Cohort 1: Sequence AEBDC (Days 1, 5, 9, 13, and 17) | Cohort 1: Sequence EADBC (Days 1, 5, 9, 13, and 17) | Cohort 1: Sequence EDACB (Days 1, 5, 9, 13, and 17) | Cohort 1: Sequence DECAB (Days 1, 5, 9, 13, and 17) | Cohort 1: Sequence BACED (Days 1, 5, 9, 13, and 17) | Cohort 1: Sequence BCADE (Days 1, 5, 9, 13, and 17) | Cohort 1: Sequence CBDAE (Days 1, 5, 9, 13, and 17) | Cohort 1: Sequence CDBEA (Days 1, 5, 9, 13, and 17) | Cohort 1: Sequence DCEBA (Days 1, 5, 9, 13, and 17) | Cohort 3: Sequence IJK (Days 1, 5, and 9) | Cohort 3: Sequence JKI (Days 1, 5, and 9) | Cohort 3: Sequence KIJ (Days 1, 5, and 9)
Started | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 5 | 5 | 5
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 2 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Treatment A: RDEA3170 capsules, 5 mg (FN24), administered in the fasted state. Treatment B: RDEA3170 capsules, 5 mg FN24, administered in the fed state (high-fat, high-calorie meal). Treatment C: RDEA3170 capsules, 10 mg (FN25), administered in the fasted state. Treatment D: RDEA3170 capsules, 10 mg FN25, administered in the fed state (high-fat, high-calorie meal). Treatment E: RDEA3170 tablets, 2.5 mg FN17, administered as 10 mg (4 × 2.5 mg), in the fasted state.
- Cohort 3 (Optional): Treatment I: RDEA3170 capsules, 10 mg (FN26), administered in the fasted state. Treatment J: RDEA3170 capsules, 10 mg FN26, administered in the fed state (high-fat, high-calorie meal).
  Treatment K: RDEA3170 tablets, 2.5 mg FN17, administered as 10 mg (4 × 2.5 mg), in the fasted state
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 3 (Optional) | Total
Number analyzed (Participants) | 20 | 15 | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35 (8.9) | 41 (12.0) | 38 (10.45)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 20 | 15 | 35
  Female | 0 | 0 | 0
Region of Enrollment [Number; unit: Participants]
  United States | 20 | 15 | 35

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax is the maximum observed concentration of a drug after administration
Time Frame: Day 1, 5, 9, 13, 17
Population: A subject in Treatment A was excluded from pharmacokinetic (PK) analysis on Day 13 following oral administration of 5 mg (FN24) capsules under the fasted condition due to a suspected dosing error. There was no evaluable PK available on Day 13 for this subject.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Groups:
- Treatment A: Verinurad capsules, 5 mg (FN24), administered in the fasted state.
- Treatment C: Verinurad capsules, 10 mg (FN25), administered in the fasted state.
- Treatment E; Treatment K: RDEA3170 tablets, 2.5 mg (FN17), administered as 10 mg (4 × 2.5 mg), in the fasted state.
- Treatment I: RDEA3170 capsules, 10 mg (FN26), administered in the fasted state.
Arm/Group | Treatment A | Treatment C | Treatment E | Treatment I | Treatment K
Number analyzed (Participants) | 19 | 20 | 20 | 15 | 15
ng/mL | 14.9 [12.5 to 17.8] | 23.4 [19.3 to 28.2] | 12.9 [11.2 to 14.9] | 14.0 [12.1 to 16.3] | 13.2 [11.2 to 15.5]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Test type: Non-Inferiority or Equivalence — The sample size is not based on formal power calculations, as this study is designed only to provide an initial assessment of the Pharmacokinetics (PK), Pharmacodynamics (PD), and safety profile of RDEA3170; Mixed Models Analysis; A mixed effect model on the natural log-transformed PK parameters Cmax, AUClast, and AUC∞ with fixed effect for treatment; Geometric Least Squares Mean Ratio = 232, 90% CI 2-sided [202 to 266]
Statistical Analysis 2: Comparison: Treatment C vs Treatment E; Test type: Non-Inferiority or Equivalence — The sample size is not based on formal power calculations, as this study is designed only to provide an initial assessment of the PK, PD, and safety profile of RDEA3170; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 181, 90% CI 2-sided [164 to 200]
Statistical Analysis 3: Comparison: Treatment I vs Treatment K; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 106, 90% CI 2-sided [91.5 to 124]

2. Primary Outcome: Time of Occurrence of Maximum Observed Concentration (Tmax)
Description: Tmax is the time of occurrence of cmax
Time Frame: Day 1, 5, 9, 13, 17
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Groups:
- Treatment B: RDEA3170 capsules, 5 mg (FN24), administered in the fed state (highfat, high-calorie meal).
- Treatment D: RDEA3170 capsules, 10 mg (FN25), administered in the fed state (high-fat, high-calorie meal)
- Treatment J: RDEA3170 capsules, 10 mg (FN26), administered in the fed state (high-fat, high-calorie meal).
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment I | Treatment J | Treatment K
Number analyzed (Participants) | 19 | 20 | 20 | 20 | 20 | 15 | 15 | 15
hr | 3.00 (2.05) [1.00 to 4.00] | 4.00 (1.69) [3.00 to 10.0] | 3.50 (1.74) [1.00 to 6.00] | 4.00 (1.05) [3.00 to 8.00] | 2.00 (1.54) [1.00 to 4.00] | 2.00 (2.71) [1.00 to 6.00] | 6.00 (2.45) [3.00 to 12.0] | 3.00 (2.66) [1.00 to 6.00]

3. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Quantifiable Last Sampling Timepoint (AUC Last)
Description: AUC last is the area under the plasma concentration time curve from zero to the last quantifiable sampling timepoint
Time Frame: Day 1, 5, 9, 13, 17
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng·hr/mL
Arm/Group | Treatment A | Treatment C | Treatment E | Treatment I | Treatment K
Number analyzed (Participants) | 19 | 20 | 20 | 15 | 15
ng·hr/mL | 91.2 [80.6 to 103] | 185 [163 to 211] | 109 [89.9 to 132] | 149 [130 to 171] | 115 [96.9 to 137]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 170, 90% CI 2-sided [147 to 195]
Statistical Analysis 2: Comparison: Treatment C vs Treatment E; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 170, 90% CI 2-sided [146 to 199]
Statistical Analysis 3: Comparison: Treatment I vs Treatment K; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 129, 90% CI 2-sided [114 to 146]

4. Primary Outcome: Area Under the Concentration-time Curve From 0 to Infinity (AUC∞)
Description: AUC 0-∞ is a meausre of total concentration from time zero to infinity
Time Frame: Day 1, 5, 9, 13, 17
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng·hr/mL
Arm/Group | Treatment A | Treatment C | Treatment E | Treatment I | Treatment K
Number analyzed (Participants) | 19 | 20 | 20 | 20 | 20
ng·hr/mL | 95.7 [84.5 to 108] | 192 [169 to 219] | 121 [97.0 to 150] | 161 [140 to 184] | 123 [103 to 146]
Statistical Analysis 1: Comparison: Treatment A vs Treatment E; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 161, 90% CI 2-sided [139 to 187]
Statistical Analysis 2: Comparison: Treatment C vs Treatment E; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 159, 90% CI 2-sided [135 to 188]
Statistical Analysis 3: Comparison: Treatment I vs Treatment K; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 131, 90% CI 2-sided [116 to 147]

5. Primary Outcome: Apparent Terminal Half-life (t1/2)
Description: t1/2 is a measure of apparent terminal half-life
Time Frame: Day 1, 5, 9, 13, 17
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: hr
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment I | Treatment J | Treatment K
Number analyzed (Participants) | 19 | 20 | 20 | 20 | 20 | 15 | 15 | 15
hr | 13.6 (2.05) [11.2 to 16.5] | 14.9 (1.69) [12.6 to 17.6] | 14.0 (1.74) [11.5 to 17.0] | 12.9 (1.05) [10.6 to 15.6] | 17.3 (1.54) [13.4 to 22.3] | 14.4 (2.71) [9.70 to 21.5] | 15.8 (2.45) [11.6 to 21.5] | 13.2 (2.66) [9.44 to 18.6]

6. Primary Outcome: Maximum Observed Plasma Concentration (Cmax): Effect of High Fat Meal on the PK of RDEA3170 Capsules
Description: Cmax is the maximum observed concentration of a drug after administration
Time Frame: Day 1, 5, 9, 13, 17
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment I | Treatment J
Number analyzed (Participants) | 19 | 20 | 20 | 20 | 15 | 15
ng/mL | 14.9 [12.5 to 17.8] | 15.0 [12.6 to 18.0] | 23.4 [19.3 to 28.2] | 23.3 [19.2 to 28.3] | 14.0 [12.1 to 16.3] | 16.3 [12.9 to 20.7]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 99.4, 90% CI 2-sided [88.3 to 112]
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 99.9, 90% CI 2-sided [85.5 to 117]
Statistical Analysis 3: Comparison: Treatment I vs Treatment J; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 116, 90% CI 2-sided [94.8 to 143]

7. Primary Outcome: AUC Last: Effect of High Fat Meal on the PK of RDEA3170 Capsules
Description: AUC last is the area under the plasma concentration time curve from zero to the last quantifiable sampling timepoint
Time Frame: Day 1, 5, 9, 13, 17
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng·hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment I | Treatment J
Number analyzed (Participants) | 19 | 20 | 20 | 20 | 15 | 15
ng·hr/mL | 91.2 [80.6 to 103] | 99.2 [86.4 to 114] | 185 [163 to 211] | 192 [171 to 216] | 149 [130 to 171] | 172 [136 to 218]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 107, 90% CI 2-sided [98.3 to 116]
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 104, 90% CI 2-sided [95.0 to 113]
Statistical Analysis 3: Comparison: Treatment I vs Treatment J; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 115, 90% CI 2-sided [95.3 to 140]

8. Primary Outcome: AUC∞: Effect of High Fat Meal on the PK of RDEA3170 Capsules
Description: AUC 0-∞ is a meausre of total concentration from time zero to infinity
Time Frame: Day 1, 5, 9, 13, 17
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ng·hr/mL
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment I | Treatment J
Number analyzed (Participants) | 19 | 20 | 20 | 20 | 15 | 15
ng·hr/mL | 95.7 [84.5 to 108] | 104 [90.5 to 119] | 192 [169 to 219] | 199 [177 to 224] | 161 [140 to 184] | 182 [142 to 233]
Statistical Analysis 1: Comparison: Treatment A vs Treatment B; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 107, 90% CI 2-sided [98.1 to 116]
Statistical Analysis 2: Comparison: Treatment C vs Treatment D; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 103, 90% CI 2-sided [94.6 to 113]
Statistical Analysis 3: Comparison: Treatment I vs Treatment J; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 2]; Mixed Models Analysis; [statistical method as in outcome 1, analysis 1]; Geometric Least Squares mean Ratio = 113, 90% CI 2-sided [93.3 to 137]

9. Secondary Outcome: Pharmacodynamics (PD) Profile of RDEA3170
Description: Serum samples were collected at the following timepoints in relation to RDEA3170 dosing: Day 1 (Cohort 1 and Cohort 3): -24, -23, -22, -21, -20, -18, -16, -14, and -12 hours prior to dosing. Days 1, 5, and 9 (Cohort 1 and Cohort 3), and Days 13 and 17 (Cohort 1 only): predose (within 30 minutes prior to dosing) and 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose. Urine samples (total catch) were collected at the following timepoints in relation to RDEA3170 dosing: Day 1 (Cohort 1 and Cohort 3): -24 to -21, -21 to -18, -18 to -12, and -12 to 0 hours predose. Days 1, 5, and 9 (Cohort 1 and Cohort 3), and Days 13 and 17 (Cohort 1 only): 0 to 3, 3 to 6, 6 to 12, and 12 to 24 hours postdose.
Time Frame: Day -1, 1, 5, 9, 13, 17
Population: A subject in Treatment A was excluded from pharmacokinetic (PK) analysis on Day 13 (but not from pharmacodynamics analysis) following oral administration of 5 mg (FN24) capsules under the fasted condition due to a suspected dosing error. There was no evaluable PK available on Day 13 for this subject.
Measure: Mean (Standard Error); unit: Percent (%) Change
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment I | Treatment J | Treatment K
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 15 | 15 | 15
Percent (%) Change
  Serum Urate Maximum % Change | -29.1 (2.05) | -40.6 (1.69) | -42.5 (1.74) | -52.3 (1.05) | -30.3 (1.54) | -35.2 (2.71) | -46.2 (2.45) | -29.3 (2.66)
  Urine Uric Acid % Change (0-24h) | 79.2 (21.6) [33.9 to 124] | 92.3 (19.0) [52.5 to 132] | 109 (27.8) [51.2 to 168] | 88.8 (13.6) [60.3 to 117] | 76.8 (14.4) [46.6 to 107] | 49.5 (8.22) [31.9 to 67.1] | 53.7 (8.56) [35.4 to 72.1] | 53.9 (10.0) [32.4 to 75.3]
  Renal Clearance of Uric Acid % Change (0-24h) | 137 (33.1) [10.9 to 14.6] | 175 (27.2) [13.9 to 17.2] | 226 (48.4) [15.3 to 20.1] | 216 (23.7) [15.1 to 20.9] | 142 (27.1) [11.7 to 15.3] | 117 (17.4) [12.0 to 16.5] | 153 (17.2) [14.4 to 19.8] | 107 (17.7) [11.6 to 15.4]
  Fractional Excretion of uric acid % Change (0-24h) | 119 (13.1) [9.82 to 13.3] | 157 (12.9) [12.0 to 15.5] | 214 (14.5) [15.0 to 18.8] | 214 (14.3) [15.0 to 18.6] | 145 (15.1) [11.1 to 14.7] | 137 (18.4) [11.2 to 15.3] | 168 (15.5) [13.5 to 17.6] | 120 (14.2) [10.5 to 14.3]

10. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events
Time Frame: 8 weeks
Population: The safety population included all participants who received any dose of investigational product.
Measure: Number; unit: Number of participants
Groups:
- Treatmnet K: RDEA3170 tablets, 2.5 mg (FN17), administered as 10 mg (4 × 2.5 mg), in the fasted state
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment I | Treatment J | Treatmnet K
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 20 | 15 | 15 | 15
Number of participants | 1 | 1 | 0 | 0 | 0 | 2 | 2 | 0

ADVERSE EVENTS:
Description: Overall number of baseline participants used to determine number of participants at risk.
Groups:
- Treatment B: Verinurad capsules, 5 mg (FN24), administered in the fed state (highfat, high-calorie meal).
- Treatment I: Verinurad capsules, 10 mg (FN26), administered in the fasted state.
- Treatment J: Verinurad capsules, 10 mg (FN26), administered in the fed state (high-fat, high-calorie meal).
- Treatment K: Verinurad tablets, 2.5 mg (FN17), administered as 10 mg (4 × 2.5 mg), in the fasted state.
Arm/Group | Treatment A | Treatment B | Treatment C | Treatment D | Treatment E | Treatment I | Treatment J | Treatment K
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/20 | 0/20 | 0/20 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 1/20 | 1/20 | 0/20 | 0/20 | 0/20 | 2/15 | 2/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=20) | Treatment B (N=20) | Treatment C (N=20) | Treatment D (N=20) | Treatment E (N=20) | Treatment I (N=15) | Treatment J (N=15) | Treatment K (N=15)
Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall submit a copy of the Publication to Sponsor for review at least 45 days prior to its proposed submission. Sponsor reserves the right to delay any such publication for an additional period of 60 days. Upon Sponsor's request, PI agrees to delete from the proposed publication any Confidential Information. PI agrees not to release any publication without the prior written permission of Sponsor.